CLINICAL TRIAL: NCT05753774
Title: Efficacy and Safety of Fecal Microbiota Transplantation in the Treatment of Functional Gastrointestinal Disorders in Children
Brief Title: Effect of Fecal Microbiota Transplantation (FMT) in Pediatric Functional Gastrointestinal Disorders
Acronym: FGIDs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biao Zou (Other)
Responsible Party: Sponsor-Investigator, Biao Zou, associate professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 63639582
Record Dates: First submitted 2023-02-11; First posted 2023-03-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: Functional Gastrointestinal Disorders;; FMT;; Safety; efficacy; efficacy
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Fecal Microbiota Transplantation; Cyproheptadine

STUDY DESIGN:
Intervention Model Description: Children with functional gastrointestinal disease were divided into two groups, one group was given FMT combined with conventional drug intervention, and the other group was given conventional drug intervention, including: probiotics and/or omeprazole, and/or cyproheptadine, and/or amitriptyline, and/or moxapride
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fecal microbiota transplantation (Active Comparator): Fecal microbiota transplantation routes include the upper digestive tract, lower digestive tract, or oral fecal microbiota transplantation capsules
  Interventions: Biological: FMT
- Conventional drug intervention (Sham Comparator): Conventional drugs include: probiotics and omeprazole, and cyproheptadine and moxapride.
  Interventions: Drug: Conventional drugs

INTERVENTIONS:
Biological: FMT — FMT is a technique in which intestinal microbiota are transferred from a healthy screened donor to a patient, with the goal being to introduce or restore a stable microbial community in the gut. FMT was given 1-3courses, 3-6 times per courses
  Other Names: fecal microbiota transplantation
  Arms: fecal microbiota transplantation
Drug: Conventional drugs — Conventional drugs include probiotics and omeprazole, and cyproheptadine and moxapride
  Other Names: cyproheptadine
  Arms: Conventional drug intervention

SUMMARY:
Safety and efficacy of FMT in Pediatric Functional Gastrointestinal Disorders

DETAILED DESCRIPTION:
The gut microbiota is critical to health and functions with a level of complexity comparable to that of an organ system. Dysbiosis, or alterations of this gut microbiota ecology, have been implicated in a number of disease states. Functional gastrointestinal disorders (FGIDs), also known as brain-intestinal interaction abnormalities, are associated with dynamic disorders, high visceral sensitivity, changes in mucosal and immune functions, changes in intestinal flora, and abnormal central nervous system regulatory functions. Fecal microbiota transplantation (FMT) is a process in which a presumed healthy and diverse microbiome is transplanted to a patient using a nasogastric tube, colonoscopy, or enema, or Fecal capsule to remodel the intestinal flora balance. At present, there are few clinical studies on the treatment of FGID in children with FMT. The investigators prospectively enrolled functional children who met the Rome IV standard, and divided them into conventional treatment group or FMT group with open choice. The efficacy of the two groups was collected and compared at different time points, and the flora of children in the FMT group before and after treatment was collected to monitor FMT-related adverse reactions

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis and classification of patients with FGIDs were in accordance with the ROME IV criteria for children

Exclusion Criteria:

* organic gastrointestinal disease (as established by medical history, blood routine, biochemistry, c-reaction protein, erythrocyte sedimentation rate, and fecal routine examinations.)
* other chronic disease
* growth failure

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
The efficacy of FMT in pediatric FGID | 4 weeks and 8 weeks
  change in Gastrointestinal Symptom Rating Scale (GSRS), validated scale of GI symptoms. The items are scored between 1 and 7, where 1 corresponds to "no discomfort at all" and 7 to "very severe discomfort" from the symptom.
self-reported severity of pain | 4 weeks and 8 weeks
  change in self-reported severity of pain is defined as at least two Faces Pain Score (Wong-Baker Pain Rating Scale;0-no hurt,10-hurts worst for pain)

SECONDARY OUTCOMES:
Change in Pittsburgh sleep quality index (PSQI) | 4 weeks and 8 weeks
  PSQI assesses sleep quality in children. A higher score indicates poorer sleep quality. The PSQI will be assessed from baseline to 1 weeks and from baseline to 1 month. PSQI is scored from 0 to 21 points. The higher the score, the worse the sleep. PSQI≥8 was poor sleep quality, and 7 was the cut-off value
Mean number of bowel movements per week | 4 weeks and 8weeks
  change in the mean number of bowel movements per week
Bristol stool scale | 4 weeks and 8 weeks
  Change in stool consistency assessed using the Bristol Stool Form Scale. The Bristol stool classification divides stool into seven categories. Types 1 and 2 indicate constipation; Types 3 and 4 are ideal for bowel movements, while types 5 to 7 indicate possible diarrhea.
Irritable bowel syndrome Symptom Severity Scale (IBS-SSS) | 4 weeks and 8 weeks
  IBS-SSS is a visual assessment scale (VAS) rating from 0 to 100, with total scores ranging from 0 to 500. Mild, moderate and severe cases are indicated by scores of 75 to 175, 175 to 300 and > 300.
gut microbial | 4 weeks and/or 8 weeks
  Fecal 16S RNA or macrogene sequencing was performed. Fecal samples were obtained from donor and recipient. The fecal samples and isolated microbiota samples were frozen immediately and underwent DNA extraction using standard methods.
Adverse events | 2 weeks , 4 weeks and 8 weeks
  All possible adverse events after FMT: fever, abdominal pain, infectious diseases and others

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Huang, Study Director — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, China